CLINICAL TRIAL: NCT01179425
Title: Sex Differences in Attentional Bias and Cognitive Functioning in Response to Stress in Marijuana-dependent Individuals
Brief Title: Sex Differences in Attentional Bias in Marijuana-dependent Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Kimber L. Price, Ph.D., Medical University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: HR# 19292
Record Dates: First submitted 2009-11-17; First posted 2010-08-11 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Marijuana Dependence
Keywords: marijuana; dependence; cognition; stress
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-marijuana dependent controls (Active Comparator)
  Interventions: Other: Cognitive stressor
- Marijuana-dependent subjects (Experimental)
  Interventions: Other: Cognitive stressor

INTERVENTIONS:
Other: Cognitive stressor — The Paced Auditory Serial Addition Task (PASAT-C), has been modified for use as a computerized laboratory-based stressor. Single digits are presented, and the patient must add each new digit to the one immediately prior to it and click on the appropriate answer. Failure to do so in the allotted time results in a noxious error sound.

SUMMARY:
The purpose of this study is to explore sex differences in cognitive functioning and responses to marijuana-related items, and to determine whether stress impacts these measures.

Hypothesis 1: Attentional bias will be greater for marijuana cues in male marijuana-dependent subjects relative to female marijuana-dependent or non-dependent male controls.

Hypothesis 2: Marijuana-dependent females will exhibit greater stress-induced changes in attentional bias and cognitive functioning than marijuana-dependent males.

DETAILED DESCRIPTION:
Ample evidence implicates both environmental cues and negative affective states in maintaining drug use or triggering relapse. However, although 'craving' is believed to drive continued drug use, it is not well understood how cognitive processes influence craving and relapse, nor how they may differ between the sexes. Therefore, the goal of this study protocol is to provide insight into sex differences in the cognitive aspects of drug craving and to assess the impact of stress on attentional bias for drug-related cues as well as on the availability of cognitive resources.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include subjects between the ages of 18-65 who meet full DSM-IV criteria for marijuana dependence and non-dependent controls.

Exclusion Criteria:

* Exclusion criteria will include medications that may affect cognitive or HPA-axis functioning
* Current depression
* Bipolar disorder
* Attention deficit hyperactivity disorder
* History of psychosis
* Suicidal or homicidal intent
* Significant cognitive deficits
* Dependence on any substance other than marijuana, nicotine, or caffeine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures will be obtained from the auditory odd-ball task: differences while viewing the marijuana vs neutral video in reaction time (msec), errors of omission (%), and errors of commission (%). | ~ 3 hours

SECONDARY OUTCOMES:
Secondary measures include subjective (craving and stress), physiological (heart rate and skin conductance), and stress hormone level (cortisol) assessments. | ~ 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kimber L Price, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Dept. of Psychiatry/Clinical Neuroscience Division, Charleston, South Carolina, United States